CLINICAL TRIAL: NCT00734929
Title: A Comparison of the Combination of Aprepitant and Dexamethasone Versus the Combination of Ondansetron and Dexamethasone for the Prevention of Postoperative Nausea and Vomiting (PONV) in Patients Undergoing Craniotomy
Brief Title: Aprepitant With Dexamethasone Versus Ondansetron With Dexamethasone for PONV Prophylaxis in Patients Having Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00001404
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; nausea; emesis; antiemetics; aprepitant; ondansetron; dexamethasone
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Aprepitant; Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aprepitant 40 mg preoperatively + dexamethasone 10 mg after induction of anesthesia
  Interventions: Drug: Aprepitant + Dexamethasone
- 2 (Active Comparator): Ondansetron 4 mg within 30 min of the end of surgery + Dexamethasone 10 mg after induction of anesthesia
  Interventions: Drug: Ondansetron + Dexamethasone

INTERVENTIONS:
Drug: Aprepitant + Dexamethasone — Aprepitant 40 mg + Dexamethasone 10 mg
  Arms: 1
Drug: Ondansetron + Dexamethasone — Ondansetron 4 mg + Dexamethasone 10 mg
  Arms: 2

SUMMARY:
We hypothesize that the combination of aprepitant with dexamethasone will provide significantly improved prophylaxis against Postoperative nausea and vomiting compared with the combination of ondansetron and dexamethasone, in patients undergoing craniotomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

A patient is eligible for inclusion in this study if all of the following criteria apply:

* Age: 18-75 years of age
* Surgery: craniotomy under general anesthesia.
* American Society of Anesthesiologists (ASA) Status: ASA: I, II, or III
* Language: Fluent in the English language
* Informed Consent: Written informed consent must be obtained.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any one or more of the following criteria apply within thirty days of patient enrollment in this clinical trial:

* Medical: Any condition that may impair a patient's ability to complete any of the study assessments or confound interpretation of results.
* Hypersensitivity: Patient has a known immediate or delayed hypersensitivity reaction or known idiosyncrasy to any of the two study medications, ondansetron, or aprepitant.
* Other Drugs: Patients should not be taking medications with known antiemetic properties (phenothiazines, butyrophenones, antihistamines), nor should they receive metoclopramide, or other antiemetics preoperatively or 12 hours before the scheduled surgical procedure.
* Pregnant or lactating females: A pregnancy test will be performed within 24 hours of entering the study for females of childbearing potential.
* Substance Abuse: Clinically significant abuse of substances (alcohol, illicit or prescribed medications) such that the patient is unable to provide informed consent or reliably complete any of the study assessments.
* Psychiatric Disease: History of a psychiatric illness that may impair the patient's ability to provide informed consent or complete any of the study assessments.
* Nausea verbal rating score (VRS): A VRS nausea score > 3 (scale 0-10) in the preoperative holding area before pretreatment with the study medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Habib, MBBCH, FRCA, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Habib AS, Keifer JC, Borel CO, White WD, Gan TJ. A comparison of the combination of aprepitant and dexamethasone versus the combination of ondansetron and dexamethasone for the prevention of postoperative nausea and vomiting in patients undergoing craniotomy. Anesth Analg. 2011 Apr;112(4):813-8. doi: 10.1213/ANE.0b013e3181ff47e2. Epub 2010 Nov 16. PMID 21081776

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at Duke University Medical Center from September 2007 to June 2009, 146 signed the consent form, 115 were randomized, 104 completed the study
Groups:
- Aprepitant: Aprepitant 40 mg preoperatively + dexamethasone 10 mg after induction of anesthesia
- Ondansetron: Ondansetron 4 mg within 30 minutes of the end of surgery + Dexamethasone 10 mg after induction of anesthesia
Period: Overall Study
Arm/Group | Aprepitant | Ondansetron
Started | 57 | 58
Completed | 51 | 53
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — No intervention/ screen fail | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant | Ondansetron | Total
Number analyzed (Participants) | 57 | 58 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 58 | 115
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13) | 48 (13) | 50 (13)
Sex/Gender, Customized [Number; unit: participants]
  Female | 34 | 30 | 64
  Male | 22 | 29 | 51
Region of Enrollment [Number; unit: participants]
  United States | 57 | 58 | 115

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Emesis
Description: Any vomiting or retching
Time Frame: 48 h
Population: ITT analysis
Measure: Number; unit: participants
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
participants | 8 | 20

2. Secondary Outcome: Incidence of Nausea
Description: operative procedure
Time Frame: Post operative procedure (OP) hours (0-2, 24, 48)
Measure: Number; unit: participants
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
participants
  0-2 hours Post OP | 27 | 27
  24 Hours Post Op | 33 | 30
  48 Hours Post Op | 35 | 32

3. Secondary Outcome: Incidence of Vomiting (Post OP)
Time Frame: Post OP (0 - 2 hours)
Measure: Number; unit: participants
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
participants | 3 | 11

4. Secondary Outcome: Incidence of Vomiting (24 Hours)
Description: Any vomiting or retching
Time Frame: 24 h
Population: ITT analysis
Measure: Number; unit: participants
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
participants | 7 | 19

5. Secondary Outcome: Use of Rescue Antiemetics (Post OP)
Time Frame: Post OP (0 - 2 hours)
Measure: Number; unit: participants
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
participants | 20 | 24

6. Secondary Outcome: Use of Rescue Antiemetics (24 Hours)
Time Frame: 24 h
Measure: Number; unit: participants
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
participants | 31 | 30

7. Secondary Outcome: Use of Rescue Antiemetics (48 Hours)
Time Frame: 48 hour
Measure: Number; unit: participants
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
participants | 33 | 32

8. Secondary Outcome: Number of Participants With a Complete Response Rate
Description: complete response rate: defined as no Postoperative nausea and vomiting (PONV) and no need for rescue antiemetics.
Time Frame: 24 hours Post OP, 48 hours Post OP
Measure: Number; unit: participants
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
participants
  24 Hours Post OP | 14 | 21
  48 Hours Post OP | 11 | 19

9. Secondary Outcome: Average Nausea Score
Description: Participants verbally rated their nausea on a scale of 0-10. 0 = No nausea, 10 = worst nausea imaginable
Time Frame: Post OP hours 0-2, 24 h, 48 h
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
units on a scale
  0-2 hours post op | 0.4 [0 to 2.8] | 0.6 [0 to 2.4]
  24 hours post op | 0.8 [0 to 3.2] | 1.3 [0 to 2.8]
  48 hours post op | 0.9 [0 to 3.2] | 1.1 [0 to 3.3]

10. Secondary Outcome: Number of Vomiting Episodes
Time Frame: 48 hours
Measure: Mean (Inter-Quartile Range); unit: vomiting episodes
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
vomiting episodes | 0 [0 to 0] | 0 [0 to 1.5]

11. Secondary Outcome: Time to First Vomiting
Time Frame: 48 h
Population: The analysis population only includes participants who had vomiting and had a complete data set
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Aprepitant + Dexamethasone: Aprepitant 40 mg preoperatively + dexamethasone 10 mg after induction of anesthesia
  Aprepitant + Dexamethasone: Aprepitant 40 mg + Dexamethasone 10 mg
- Ondansetron + Dexamethasone: Ondansetron 4 mg within 30 min of the end of surgery + Dexamethasone 10 mg after induction of anesthesia
  Ondansetron + Dexamethasone: Ondansetron 4 mg + Dexamethasone 10 mg
Arm/Group | Aprepitant + Dexamethasone | Ondansetron + Dexamethasone
Number analyzed (Participants) | 6 | 19
hours | 13.5 [0.5 to 28.9] | 2 [0.5 to 19.3]

12. Secondary Outcome: Number of Participants Who Rated Their Satisfaction With Antiemetic Management as "Very Satisfied"
Description: Participants rated their satisfaction with antiemetic management on a 5 points scale: very satisfied, somewhat satisfied, neither satisfied nor dissatisfied, somewhat dissatisfied, very dissatisfied)
Time Frame: 48 hour
Measure: Number; unit: participants
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 51 | 53
participants | 36 | 32

ADVERSE EVENTS:
Arm/Group | Aprepitant | Ondansetron
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/53
Other Adverse Events (participants affected / at risk) | 0/51 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No